CLINICAL TRIAL: NCT00720811
Title: Assessment of Use of Rapid Diagnostic Testing in the Context of Home Management With ACTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: Makerere University (Other); Ministry of Health, Uganda (Other Government); Navrongo Health Research Centre, Ghana (Other); National Malaria Research and Training Centre, Burkina Faso (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A60487
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Malaria; Pneumonia
Keywords: Malaria ACT; Rapid; Diagnosis; Community; health; worker; Artemesinin; based; Combination; Therapy; Anti Malarial; Treatment; antibiotics
MeSH Terms: conditions — Malaria; Pneumonia; Fasting; Disease | interventions — Artemether, Lumefantrine Drug Combination; Amoxicillin; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT, antibiotic, paracetamol (Experimental): CHWs will test children with acute febrile illness for malaria using RDTs, and for pneumonia by counting their respiratory rate with RRTs. Treatment will then be provided on the basis of the test results, in line with national guidelines. Children with a positive RDT will receive artemether-lumefantrine in Burkina Faso and Uganda, and artesunate-amodiaquine in Ghana. Children with a cough and a high respiratory rate will receive amoxicillin in Ghana and Uganda, and cotrimoxazole in Burkina Faso. Additionally, paracetamol (PCT) will be provided to all children with an axillary temperature > 38.5°C.
  Interventions: Drug: Artemether-lumefantrine combination; Drug: amoxycillin; Drug: paracetamol; Device: malaria rapid diagnostic test, respiratory rate timer
- Presumptive fever management (No Intervention): Presumptive treatment of malaria with ACTs. No antibiotic treatment available
  Interventions: Drug: Artemether-lumefantrine combination

INTERVENTIONS:
Drug: Artemether-lumefantrine combination — 20/120mg Artemether-lumefantrine 4-35 months: 1 tablet twice daily for 3 days; 36-59 months: 2 tablets twice daily for 3 days
  Other Names: Coartem
  Arms: ACT, antibiotic, paracetamol
Drug: amoxycillin — amoxycillin 250mg tab 4-12 months: 1/2x2; 13-35 months: 1x2; 36-59 months: 11/2x2
  Arms: ACT, antibiotic, paracetamol
Drug: paracetamol — paracetamol 500mg tablet <36months: 1/4x4 for 2 days; 36-59months: 1/2x4 for 2 days
  Arms: ACT, antibiotic, paracetamol
Device: malaria rapid diagnostic test, respiratory rate timer — malaria dipstick, and breath timer
  Arms: ACT, antibiotic, paracetamol
Drug: Artemether-lumefantrine combination — 20/120mg tablet arthermether-lumefantrine 4-35months: 1x2; 36-59months: 2x2
  Arms: Presumptive fever management

SUMMARY:
This study is to assess the value of incorporating a malaria RDT based strategy in HMM. The primary activity of the study wil be a two armed cluster randomised trial in two study sites in Uganda, one in Ghana and one in Burkina Faso. One of the Uganda sites is highly endemic and the other meso-endemic for malaria. In one arm the children will be treated presumptively for malaria with ACT (control arm) and the other arm the children will receive ACT only when they have a positive RDT result (implementation arm). The children in the implementation arm will also receive antibiotics if they have a raised respiratory rate. The primary outcome will be the recovery rate in the intervention arm compared to that of the control arm on Day 3. In addition, an acceptability assessment of RDTs in the community will be undertaken both before and after the intervention trial and a cost-effectiveness analysis of the RDT strategy will also be completed. For a sub-sample, microscopy slides will also be taken on Day 0 to demonstrate comparable levels of endemicity in control and intervention groups. These activities will be carried out over a two year period.

DETAILED DESCRIPTION:
This is an open, cluster randomised multicentre two arm trial in the three countries of Burkina Faso, Ghana and Uganda. Clusters are villages (catchment populations) of individual community health workers (CHWs). Within the study areas, clusters that are more than 5 km from a designate health facility where CHWs referred cases for special care will be excluded. A cluster randomized design was chosen over an individually randomized design to reduce contamination, facilitate supervision, reduce costs, and to ensure that the CHWs maintained the correct treatments based on the tests in the Intervention arm and the presumptive treatment in the Control arm.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4-59 months of age with a history of fever in the last 24 hours presenting to the community medicine distributor

Exclusion Criteria:

* Children classified as having severe illness according to IMCI guidelines. Children suffering from Chronic disease(s), those with reported anti malarial or antibiotic treatment (intervention) arm in previous two weeks and those whose caregivers refuse to consent to participate

Ages: 4 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6456 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Recovery rate from fever at Day 3 | Day 3

SECONDARY OUTCOMES:
use of antimalarial and antibiotic drugs by community health workers | After patient enrollment
Recovery rate from fever at Day 7 | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Francis Bajunirwe, MBChB PhD, Study Director — Mbarara University of Science and Technology; George Pariyo, MB ChB, PhD, Study Director — Makerere University; James Tibenderana, MB ChB, PhD, Principal Investigator — Malaria Consortium; Alfred Tiono, PhD, Principal Investigator — National Malaria Research and Training Center, Burkina Faso; Thomas Anyorigiya, MSc, Principal Investigator — Navrongo Health Research Centre, Ghana
Locations (4):
- Sapone Site, Saponé, Burkina Faso
- Kassena Nankana Site, Kassane, Ghana
- Uganda (2):
  - Iganga Site, Iganga
  - Mbarara Site, Mbarara